CLINICAL TRIAL: NCT03783208
Title: Intrauterine G-CSF Administration in Recurrent Implantation Failure
Brief Title: Intrauterine G-CSF Administration in RIF
Acronym: G-CSF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gurgan Clinic (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20182
Record Dates: First submitted 2018-12-19; First posted 2018-12-20 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Infertility
Keywords: Endometrium; G-CSF; Recurrent implantation failure
MeSH Terms: conditions — Infertility | interventions — Granulocyte Colony-Stimulating Factor; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- G-CSF (Experimental): Patients in the G-CSF group will receive G-CSF once a day on hCG day, before hCG injection. The procedure involved the administration of G-CSF through slow infusion into the endometrial cavity using a soft embryo transfer catheter.
  Interventions: Drug: G-CSF
- Control group (Placebo Comparator): Normal saline of 1 mL was infused into the endometrial cavity in the same way in patients in the control group
  Interventions: Other: Saline

INTERVENTIONS:
Drug: G-CSF — Slow infusion of G-CSF into the endometrial cavity using a soft embryo transfer catheter.
  Other Names: Leucostim
  Arms: G-CSF
Other: Saline — Slow infusion of saline into the endometrial cavity using a soft embryo transfer catheter.
  Arms: Control group

SUMMARY:
Aim of this study is to investigate the effects of intrauterine G-CSF on endometrial thickness, clinical pregnancy rate and live birth rate in a recurrent implantation failure (RIF) group

DETAILED DESCRIPTION:
This study was designed as a prospective randomized controlled trial with the involvement of 200 RIF group patients.The procedure will perform by administering 30 mIU of Leucostim®(Filgrastim [G-CSF] 30mIU/mL; DEM Medical, Dong-A; South Korea) through slow infusion into the endometrial cavity using a soft embryo transfer catheter. Normal saline of 1 mL will be infused into the endometrial cavity in the same way in the control group. The standard ICSI procedure will use for all patients, and fresh cycle embryos will be transferred on the third or fifth day.

ELIGIBILITY:
Inclusion Criteria:

* Women under the age of 40 who met the RIF definition
* Follicle-stimulating hormone (FSH) levels were <15 IU/mL

Exclusion Criteria:

* Patients with congenital uterine anomalies
* Patients with Asherman's syndrome
* Patients with uterine cavity distorted by myoma or endometrial polyps
* Patients with confirmed endometriosis or endometrioma
* Patients for whom G-CSF was contraindicated (active infections, kidney disease, sickle cell anemia, malignancies, chronic neutropenia)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female participants
Enrollment: 157 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 1month
  Gestational sac in USG per embryo transfer

SECONDARY OUTCOMES:
Endometrial thickness | 1month
  Measurement of endometrial thickness as millimeter

CONTACTS AND LOCATIONS:
Overall Officials: Ziya Kalem, MD, Principal Investigator — Gurgan Clinic IVF and Women Health Center
Locations (1):
- Gurgan Clinic IVF and Women Health Center, Ankara, Cankaya, Turkey (Türkiye)